CLINICAL TRIAL: NCT03979066
Title: A Phase 2, Open-Label, Multicenter, Randomized Study Evaluating NEOadjuvant Immunotherapy Based Combinations in Patients With Resectable PANCreatic Ductal Adenocarcinoma
Brief Title: Study Evaluating NEOadjuvant Immunotherapy in Resectable PANCreatic Ductal Adenocarcinoma
Acronym: NEOiPANC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Loss of funding
Sponsor: Gulam Manji (Other)
Collaborators: Genentech, Inc. (Industry); Halozyme Therapeutics (Industry)
Responsible Party: Sponsor-Investigator, Gulam Manji, Assistant Professor of Medicine at Columbia University Medical Center, Columbia University
Organization: Columbia University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAS1908
Record Dates: First submitted 2019-06-06; First posted 2019-06-07 (Actual); Results first posted 2020-12-23 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Pancreatic Ductal Adenocarcinoma
Keywords: Neoadjuvant therapy; PEGPH20; Atezolizumab; Columbia; Pancreatic Ductal Adenocarcinoma
MeSH Terms: interventions — atezolizumab; PEGPH20

STUDY DESIGN:
Intervention Model Description: Randomized phase 2 trial for a total of 20 patients per cohort
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Atezolizumab (Active Comparator): Atezolizumab 840mg IV every 2 weeks for 2 doses prior to surgery and 4 doses after surgery.
  Interventions: Drug: Atezolizumab
- Atezolizumab in combination with PEGPH20 (Experimental): Atezolizumab 840mg IV every 2 weeks for 2 doses prior to surgery and 4 doses after surgery in combination with PEGPH20 3ug/kg IV twice weekly for 3 weeks prior to surgery and once weekly for 3 weeks (of 28 day cycle) for two cycles after surgery.
  Interventions: Drug: Atezolizumab; Drug: PEGPH20

INTERVENTIONS:
Drug: Atezolizumab — 840mg IV every 2 weeks for 2 doses prior to surgery and 4 doses after surgery.
  Other Names: Tecentriq
Drug: PEGPH20 — PEGPH20 3ug/kg IV twice weekly for 3 weeks prior to surgery and once weekly for 3 weeks (of 28 day cycle) for two cycles after surgery.
  Other Names: pegvorhyaluronidase alfa
  Arms: Atezolizumab in combination with PEGPH20

SUMMARY:
The purpose of this study is to determine if study treatment with atezolizumab and PEGPH20 given before and after surgery, followed by chemotherapy is safe and if it can further increase the immune response against the tumor rather than increase the chance of cure.

DETAILED DESCRIPTION:
Presently, surgical resection offers the only therapeutic means of cure. However only 15%-20% of patients are found to have resectable disease at time of initial diagnosis. Of the patients who undergo curative surgery, most will relapse and eventually succumb to the disease. 5-year survival rates for node-negative and -positive disease at time of pancreatic duodenectomy are 25%-30% and 10%, respectively.

Although early phase trials have not offered great success in the metastatic setting for patients with pancreas adenocarcinoma (PDA), interim analysis of a multicenter, phase 1 trial with durvalumab presented at European Society for Medical Oncology (ESMO) indicated a disease control rate of 21%. As mentioned previously, PD-L1 expression correlates with poor prognosis and decreased CD4+ and CD8+ T cell infiltration within the tumor. Targeting PD-L1 in the micrometastatic setting (resectable disease), when robust mature immunosuppressive pathways may not have yet formed, may be the optimum time to investigate anti-PD-L1 therapy. This arm of the study aims to test if atezolizumab is able to modulate CD8+ T-cell infiltration compared to historical matched controls. As a secondary endpoint we will also evaluate how clinical outcomes compare to matched historical controls.

Neoplastic, immune, and stromal cells within PDA reside in a highly dense desmoplastic environment composed of an extracellular matrix of which hyaluronidase (HA) is an abundant component. HA is a linear glycosaminoglycan and an integral component of not only PDA tumors, but has also been shown to accumulate in many solid tumors and is associated with a poor prognosis and increased immunosuppression. In a preclinical autochthonous mouse model of PDA, Sunil Hingorani's group demonstrated that the interstitial fluid pressures were unusually high within tumors that exhibited a high HA content. Furthermore, high HA tumors contained low vascularity, which compromised delivery of chemotherapeutic agents, such as gemcitabine. Mice treated with hyaluronidase resulted in decreased HA content and microvasculature re-expansion within tumors which led to a survival benefit. These preclinical studies led to early phase clinical studies in metastatic PDA where addition of PEGPH20 to gemcitabine and nab-paclitaxel (GA) in a randomized phase 2 study demonstrated a survival benefit in patients with HA-high tumors. The objective response rate for patients who were treated with a combination of PEGPH20 and GA compared to GA alone was 45% versus 31%, respectively, and the median overall survival was 11.5 versus 8.5 months, respectively (hazard ratio (HR), 0.96; 95% Confidence Interval (CI), 0.57 to 1.61). A large phase 3 randomized clinical trial in the high HA stage IV PDA population in the first line setting is ongoing.

PDA likely invokes multiple immune evading mechanisms which result in its aggressive behavior; it is expected that multiple agents will likely be needed to develop effective therapies. One such rationale is the combination of PEGPH20 and immune checkpoint blockade to allow increased cytotoxic T-cell infiltration by increasing vascular permeability and decreasing interstitial pressure. In a breast cancer preclinical model, PEGPH20 resulted in an increase accumulation of CD8+ tumor-infiltrating lymphocytes (TIL) by 176% (p=0.0025) and improved tumor growth inhibition by 38% relative to anti-PD-L1 alone (86% vs 62.4%, p=0.0024). Other preclinical studies are also demonstrating increased CD8+ T-cell infiltration with addition of PEGPH20 and improved tumor control in combination with immune checkpoint blockade. These and other preclinical studies suggest that this combination is worth pursuing in patients with resectable PDA. The combination is hoped to increase CD8+ T-cell infiltration within the primary tumor for improved immune mediated cytotoxicity and decreased interstitial pressure to allow improved surgical resections. Hypothetically, the combination should also be effective in foci of micrometastasis, where the tumor microenvironment (TME) may not be as mature.

Identified risks for PEGPH20 include musculoskeletal events (MSEs), infusion-related reactions (IRRs), and thromboembolic (TE) events.

ELIGIBILITY:
Inclusion Criteria:

* Histological or pathological confirmation of pancreatic adenocarcinoma Cytologic or histologic proof of PDA needs to be verified by the treating institution pathologist either from the initial diagnostic biopsy, or from the required pre treatment biopsy and prior to initiation of any study-related therapy
* Extent of disease. Stage 1 or 2 PDA and patient deemed a surgical candidate by the PI in consultation with the designated site radiologist and surgeon at the treating institution
* No prior surgical, systemic or radiotherapy for PDA.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Minimum age of at least 18 years.
* Adequate hematological and end-organ function, defined by laboratory test results, obtained within 14 days prior to initiation of study treatment:
* Tumor accessible for fresh biopsy
* Women of child-bearing potential must have a negative serum pregnancy test at screening and must agree to use two forms of effective contraception from the time of the negative pregnancy test and for a minimum of 5 months after the last dose of study drug. Women will be considered not of child-bearing potential if amenorrheic at least for one year or have undergone surgical sterilization.
* Fertile men must agree to use an effective method of birth control during the study and for up to 5 months after the last dose of study drug.
* Willingness and ability to provide written informed consent prior to any study-related procedures and to comply with all study requirements.
* Able to comply with the study protocol, in the investigator's judgment.

Exclusion Criteria:

* Prior treatment with T-cell co-stimulating or immune checkpoint blockade therapies, including but not limited to anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies.
* Patients who are receiving any other investigational agents concurrently.
* Concomitant treatment with other anti-neoplastic agents (hormonal therapy acceptable).
* Uncontrolled pleural effusion, pericardial effusion, or ascites.
* Patient receiving therapeutic doses of anticoagulation.
* Uncontrolled hypercalcemia or symptomatic hypercalcemia requiring continued use of bisphosphonate therapy.
* Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, or multiple sclerosis, with the following exceptions:
* Patients with a history of autoimmune-related hypothyroidism who are on thyroid replacement hormone are eligible for the study.
* Patients with controlled Type 1 diabetes mellitus who are on a stable insulin regimen are eligible for the study.
* Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:
* Rash must cover < 10% of body surface area.
* Disease is well controlled at baseline and requires only low-potency topical corticosteroids.
* No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months.
* History of idiopathic pulmonary fibrosis, interstitial lung disease, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan
* History of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Positive HIV test at screening or at any time prior to screening. Patients without a prior positive HIV test result will undergo an HIV test at screening, unless not permitted per local regulations.
* Active hepatitis B virus (HBV) infection (chronic or acute)
* Active hepatitis C virus (HCV) infection
* Known active tuberculosis.
* Severe infection within 4 weeks prior to initiation of study treatment
* Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment except for biliary tract infection due to bile duct obstruction from the pancreas mass. Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.
* Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 12 months prior to initiation of study treatment, seizure disorder, uncontrolled hypertension, or unstable arrhythmia or unstable angina within 3 months prior to initiation of study treatment.
* Grade ≥3 hemorrhage or bleeding event within 28 days prior to initiation of study treatment.
* Prior autologous stem cell, allogeneic stem cell, or solid organ transplantation.
* History of malignancy other than PDA within 2 years prior to screening, with the exception of those with a negligible risk of metastasis or death (e.g., 5-year overall survival of > 90%), such as adequately treated carcinoma in situ of the cervix, nonmelanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer. Patients with history of prior malignancies should have risk of recurrence within 3 years after screening to be less than 90% (to be discussed with the PI for final determination of eligibility).
* Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during treatment with atezolizumab or within 5 months after the last dose of atezolizumab.
* History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins.
* Known hypersensitivity to Chinese hamster ovary cell products or recombinant human antibodies.
* Known allergy or hypersensitivity to any of the study drugs or any of their excipients.
* Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2) within 4 weeks or five half-lives of the drug (whichever is longer) prior to initiation of study treatment.
* Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor alpha agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during the course of the study, with the following exceptions:
* Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study if receiving equivalent to less than 10mg of prednisone daily.
* Patients who received a one-time pulse dose of systemic immunosuppressant medication are eligible for the study after approval from the PI has been obtained.
* Inability to swallow medication or malabsorption condition that would alter the absorption of orally administered medications.
* Pregnant women are excluded from this study because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with these agents and breastfeeding should be discontinued.
* Major surgical procedure or significant traumatic injury within 14 days of initiating study.
* Previous radiotherapy to 25% or more of the bone marrow.
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications in the opinion of the treating investigator.
* Considered ineligible to receive full standard dose modified FOLFIRINOX therapy in the adjuvant setting.
* Peripheral neuropathy > Grade 1
* History of allergy or hypersensitivity to oxaliplatin, irinotecan, leucovorin, fluorouracil, pegfilgrastim, or any excipients.
* History of Gilbert's disease or known genotype UGT1A1 * 28/* 28.6.2.35 Inflammatory disease of the colon or rectum, or severe uncontrolled diarrhea.

Exclusion Criteria for PEGPH20-Containing Arm Patients who meet any of the following criteria will be excluded from the PEGPH20- containing arm:

* History of transient ischemic attack requiring intervention or treatment, carotid artery disease requiring interventions or treatment, of cerebrovascular accident
* Evidence of deep vein thrombosis (DVT), pulmonary embolism, or other thromboembolic event at screening, except:
* Superficial vein thrombosis
* Visceral or splanchnic vein thrombosis if the thrombosis is at a location near the site of underlying pancreatic ductal adenocarcinoma (PDAC) which may contribute to the etiology of the thrombus
* Treatment with megestrol acetate within 14 days prior to initiation of study treatment
* Unable to use low-molecular-weight heparin

Criteria to initiate chemotherapy

* Full recovery from surgery and subject able to receive chemotherapy.
* Subjects who have evidence of recurrent disease prior to initiation of chemotherapy will need to undergo biopsy to prove disease recurrence if deemed safe.
* Hematological: laboratory test results within protocol defined safety limits

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2019-11-03 (Actual); Study Completion 2019-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gulam Manji, MD, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant was enrolled but was not randomized, as the participant was determined to be a screen failure.
Period: Overall Study
Arm/Group | Atezolizumab | Atezolizumab in Combination With PEGPH20
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: One participant enrolled into the study. That participant was determined to be a screen failure. Data was not collected and therefore there is no data to analyze.
Groups:
- Total: Total of all reporting groups
Arm/Group | Atezolizumab | Atezolizumab in Combination With PEGPH20 | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Race (NIH/OMB)
Region of Enrollment
Study-Specific Baseline Measure

OUTCOME MEASURES:

1. Primary Outcome: Change in the Number of CD8+ T Cells Within the Tumor
Description: The change in number of intratumoral CD8+ T-cells the at time of surgery between treatment arm(s) compared to the atezolizumab arm. The CD8+ T-cell count within the tumor with neoadjuvant atezolizumab vs atezolizumab + PEGPH20 at the time of surgery will be reported using means and standard deviations by group and will be compared using a twosample T-test. If the data are not normally distributed, non-parametric models such as the Wilcoxon Rank Sum test will be used. Moreover, the distribution of CD8+ T-cell count by treatment arm will be assessed using box plots, histograms, and q-q plots.
Time Frame: At time of surgery (approximately 3 weeks)
Population: as for baseline characteristics
Arm/Group | Atezolizumab | Atezolizumab in Combination With PEGPH20
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: 18-Month Survival Rate
Description: To estimate the 18-month survival rate in patients treated with atezolizumab vs atezolizumab + PEGPH20 followed by surgery and adjuvant therapy.
Time Frame: 18 Months
Population: as for baseline characteristics
Arm/Group | Atezolizumab | Atezolizumab in Combination With PEGPH20
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Overall Survival
Description: To estimate the overall survival in patients treated with atezolizumab vs atezolizumab + PEGPH20 followed by surgery and adjuvant therapy.
Time Frame: Up to 5 years
Population: as for baseline characteristics
Arm/Group | Atezolizumab | Atezolizumab in Combination With PEGPH20
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: R0 Resection Rate
Description: To determine the R0 resection rates with atezolizumab vs atezolizumab + PEGPH20 administered in the neoadjuvant setting. R0 resection rate is defined by the proportion of patients in whom an R0 resection was achieved during surgery. R0 resection is defined by complete removal of macroscopic tumor which contains negative microscopic surgical margins. The R0 resection rate will be estimated by the number of patients in whom R0 resection was performed divided by total number of patients in each study arm. The R0 resection rate will be reported along with the exact 95% confidence interval. The investigators will compare the R0 resection rates using Fisher's exact test.
Time Frame: At time of surgery (approximately 3 weeks)
Population: One participant enrolled in the study. That participant was determined to be a screen failure. Data was not collected and therefore there is no data to analyze.
Arm/Group | Atezolizumab | Atezolizumab in Combination With PEGPH20
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Incidence of Treatment-Emergent Adverse Events
Description: To determine the safety profile with atezolizumab vs atezolizumab + PEGPH20 or other therapies followed by surgery and adjuvant therapy. The frequency and count of grade 3 or higher adverse events will be reported by treatment group. The maximum grade for each type of adverse event will also be reported.
Time Frame: Cycle 1 through 28 days after adjuvant chemotherapy period
Population: as for baseline characteristics
Arm/Group | Atezolizumab | Atezolizumab in Combination With PEGPH20
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: One participant enrolled into the study. That participant was determined to be a screen failure. Data was not collected and therefore there is no data to analyze.
Arm/Group | Atezolizumab | Atezolizumab in Combination With PEGPH20
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-13): https://cdn.clinicaltrials.gov/large-docs/66/NCT03979066/Prot_SAP_000.pdf